CLINICAL TRIAL: NCT03315234
Title: Correlation of Genetic Polymorphisms and Clinical Parameters With the Complexity of Coronary Artery Disease in the Greek Population
Brief Title: Correlation of Genetic Polymorphisms and Clinical Parameters With the Complexity of Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: LABNET IAE - Private Reference Diagnostic Laboratory (Unknown)
Responsible Party: Principal Investigator, Georgios P Rampidis, MD, MSc, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: CIP_PhD Rampidis Georgios_1.1
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Cardiovascular Risk Factor; Coronary Arteriosclerosis
Keywords: SYNTAX score; Coronary Atherosclerosis; Coronary Artery Disease; SNPs; Genetics; Genetic Risk Score; Personalized Medicine
MeSH Terms: conditions — Coronary Artery Disease; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA will be extracted from obtained subject blood samples at the AHEPA University General Hospital of Thessaloniki. DNAs will be labeled by anonymized subject ID # (de-identified), and shipped to LABNET IAE - Private Reference Diagnostic Laboratory for genotyping and genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SYNTAX score = 0: Patients with nonobstructive CAD (≤50 % diameter stenosis)
  Interventions: Genetic: SNPs associated with CAD
- 0 < SYNTAX score < 23: Low SYNTAX group
  Interventions: Genetic: SNPs associated with CAD
- SYNTAX score ≥ 23: Intermediate-High SYNTAX group
  Interventions: Genetic: SNPs associated with CAD

INTERVENTIONS:
Genetic: SNPs associated with CAD — Genotyping will be carried out by Real-Time PCR

SUMMARY:
The purpose of the research project is to investigate the potential association of 6 genetic polymorphisms with the complexity and the severity of coronary artery disease (SYNTAX score). The aim of the study is to combine genetic, clinical and laboratory data in order to create a prognostic tool that will enable an individualized therapeutic patient approach.

DETAILED DESCRIPTION:
This study focus on the prediction of future risk of cardiovascular events, assessing the severity and complexity of coronary artery disease by incorporating genetic information into the SYNTAX score and providing personalized therapeutic guidance to patients. The ultimate goal of the study would be to identify, design and develop a panel of genetic markers that in combination with clinical and angiographic information will be a reliable tool for predicting cardiovascular risk for future adverse events. Clinical and genetic patient information are systematically collected in a fashion that will enable also retrospective evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes
2. Patients giving voluntary written consent to participate in the study
3. Male or female patients between 18 years to 90 years at entry
4. Patients without previous history of CAD

Exclusion Criteria:

1. Patients < 18 years old and > 90 years old at time of coronary angiography
2. Patients with a previous history of CAD
3. Cardiac Arrest at admission
4. Patients with serious concurrent disease and life expectancy of < 1 year
5. Patients who refuse to give written consent for participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 18 years to 90 years at entry, of both genders, who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes will be studied
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between genetic risk variants and the SYNTAX score [All-comers population] | 12 months
  The investigators will evaluate the effects of 6 known genetic variants associated with risk of Coronary Artery Disease on the extend and severity of coronary atherosclerosis [as assessed by the SYNTAX score] in patients with significant CAD on coronary angiography, both individually and combined in a Genetic Risk Score

SECONDARY OUTCOMES:
MACCEs | 12 months
  Cardiovascular death, myocardial infarction, stent thrombosis, any re-intervention and stroke
Predictive value of combining a Genetic Risk Score & SYNTAX score for the prediction of 1-year MACCEs | 12 months
  A Genetic Risk Score will be calculated as the weighted sum of alleles of 6 single nucleotide polymorphisms previously associated with CAD [The GRS will be constructed by summing the number of risk alleles (0/1/2) for each of the 6 SNPs weighted by their estimated effect sizes].
  SYNTAX score is a coronary lesion complexity scoring system and represented by a single number.
Ankle-Brachial Index | At hospital admission
  A tool for diagnosing peripheral artery disease but also an indicator of systemic atherosclerosis [represented by a single number]
Left Ventricular Ejection Fraction | At hospital admission & 12 months after discharge from hospital
  LVEF [%] as assessed by echocardiography
Neutrophil to Lymphocyte Ratio | At hospital admission
  NLR [represented by a single number]
Red Cell Distribution Width | At hospital admission
  RDW [%]
Mean Platelet Volume | At hospital admission
  MPV [fL]
Glomerular Filtration Rate | At hospital admission
  GFR as assessed by CKD-EPI formula [mL/min/1.73m²]
High Density Lipoprotein | At hospital admission
  HDL [mg/dL]

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Rampidis, MD, MSc, Principal Investigator — AHEPA University Hospital, 1st Cardiology Department - PhD candidate; Georgios Sianos, MD, PhD, FESC, Principal Investigator — AHEPA University Hospital, 1st Cardiology Department - PhD Supervisor 1; Charalambos Karvounis, MD, PhD, Principal Investigator — AHEPA University Hospital, 1st Cardiology Department, Director - PhD Supervisor 2; Ioannis Vizirianakis, PharmD, PhD, Principal Investigator — Aristotle University of Thessaloniki, School of Pharmacy - PhD Supervisor 3
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Knowles JW, Zarafshar S, Pavlovic A, Goldstein BA, Tsai S, Li J, McConnell MV, Absher D, Ashley EA, Kiernan M, Ioannidis JPA, Assimes TL. Impact of a Genetic Risk Score for Coronary Artery Disease on Reducing Cardiovascular Risk: A Pilot Randomized Controlled Study. Front Cardiovasc Med. 2017 Aug 14;4:53. doi: 10.3389/fcvm.2017.00053. eCollection 2017. PMID 28856136
- [Background] Howson JMM, Zhao W, Barnes DR, Ho WK, Young R, Paul DS, Waite LL, Freitag DF, Fauman EB, Salfati EL, Sun BB, Eicher JD, Johnson AD, Sheu WHH, Nielsen SF, Lin WY, Surendran P, Malarstig A, Wilk JB, Tybjaerg-Hansen A, Rasmussen KL, Kamstrup PR, Deloukas P, Erdmann J, Kathiresan S, Samani NJ, Schunkert H, Watkins H; CARDIoGRAMplusC4D; Do R, Rader DJ, Johnson JA, Hazen SL, Quyyumi AA, Spertus JA, Pepine CJ, Franceschini N, Justice A, Reiner AP, Buyske S, Hindorff LA, Carty CL, North KE, Kooperberg C, Boerwinkle E, Young K, Graff M, Peters U, Absher D, Hsiung CA, Lee WJ, Taylor KD, Chen YH, Lee IT, Guo X, Chung RH, Hung YJ, Rotter JI, Juang JJ, Quertermous T, Wang TD, Rasheed A, Frossard P, Alam DS, Majumder AAS, Di Angelantonio E, Chowdhury R; EPIC-CVD; Chen YI, Nordestgaard BG, Assimes TL, Danesh J, Butterworth AS, Saleheen D. Fifteen new risk loci for coronary artery disease highlight arterial-wall-specific mechanisms. Nat Genet. 2017 Jul;49(7):1113-1119. doi: 10.1038/ng.3874. Epub 2017 May 22. PMID 28530674
- [Background] Assimes TL, Roberts R. Genetics: Implications for Prevention and Management of Coronary Artery Disease. J Am Coll Cardiol. 2016 Dec 27;68(25):2797-2818. doi: 10.1016/j.jacc.2016.10.039. PMID 28007143
- [Background] Vizirianakis IS, Fatouros DG. Personalized nanomedicine: paving the way to the practical clinical utility of genomics and nanotechnology advancements. Adv Drug Deliv Rev. 2012 Oct;64(13):1359-62. doi: 10.1016/j.addr.2012.09.034. Epub 2012 Sep 13. No abstract available. PMID 22983333
- [Background] Rampidis GP, Benetos G, Benz DC, Giannopoulos AA, Buechel RR. A guide for Gensini Score calculation. Atherosclerosis. 2019 Aug;287:181-183. doi: 10.1016/j.atherosclerosis.2019.05.012. Epub 2019 May 10. No abstract available. PMID 31104809
- Available data/document: Clinical Study Report: NCT03150680 — https://clinicaltrials.gov/ct2/show/NCT03150680 — GESS trial [ClinicalTrials.gov Identifier: NCT03150680] was designed exclusively based on the protocol of the study "Correlation of Genetic Polymorphisms and Clinical Parameters With the Complexity of Coronary Artery Disease" [CIP_PhD Rampidis Georgios_1.1]